CLINICAL TRIAL: NCT01612988
Title: Phase II Salvage Treatment With Bendamustine, Ofatumumab and MethylPrednisolone (BOMP) in Relapsed B-cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: Treatment With Bendamustine, Ofatumumab and MethylPrednisolone in Relapsed B-CLL
Acronym: BOMP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Other drugs others studies
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICLL01 BOMP
Record Dates: First submitted 2012-05-30; First posted 2012-06-06 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: B-cell Chronic Lymphocytic Leukemia (B-CLL)
Keywords: B-cell chronic lymphocytic leukemia; relapse; Bendamustine; Ofatumumab; Méthylprednisolone
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy BOMP (Experimental): Bendamustine, Ofatumumab and Methylprednisolone prephase and a maximum of 6 cycles every 4 weeks
  Interventions: Drug: BOMP

INTERVENTIONS:
Drug: BOMP — Day-8 OMB prephase:
  Ofatumumab 300 mg IV day -8 Methylprednisolone 100 mg TD IV day -8
  BOMP cycle 1 and 2 :
  Ofatumumab 1000 mg IV day 1 and day 15 Bendamustine 70mg IV day 2 and ady 3 Methylprednisolone 1000 mg/m² IV day 1, 2 and 3 Methylprednisolone 100 mg TD IV day 15
  BOMP cycle 3 to 6 :
  Ofatumumab 1000 mg IV day 1 Bendamustine 70mg IV day 2 and day 3 Methylprednisolone 1000 mg/m² IV day 1, 2 and 3

SUMMARY:
ICLL01 The BOMP trial: Phase II study of salvage treatment with Bendamustine, Ofatumumab and MethylPrednisolone (BOMP) in relapsed B-cell chronic lymphocytic leukemia (B-CLL).

A study of the GOELAMS / GCFLLC-MW intergroup

DETAILED DESCRIPTION:
Available datas suggest that a combination of bendamustine, ofatumumab and high dose steroids (the BOMP regimen) appears meaningful and likely to induce a high response rate in patients with relapsed CLL, including those who have relapsed after modern 1st line immuno-chemotherapy combinations and those who are fludarabine-refractory. The BOMP trial will address the complete response rate as its main objective. The results of bendamustine and rituximab CLL2M trial will serve of a comparator for the BOMP trial. Among secondary objectives, an extensive study of the p53 pathway (deletion 17p, TP53 mutational status and p53 function) will be performed and its impact on response and survival will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years and < 80 years
2. Diagnosis of CLL according IWCLL 2008 criteria and fulfilling a Matutes- Moreau score ≥ 4
3. Relapsed or refractory CLL stage A, B or C with active disease requiring therapy according to IWCLL 2008 criteria
4. Relapse or refractory after 1 to 3 previous lines including at least one line with fludarabine
5. ECOG Performance status and general condition.

   * ECOG Performance status ≤ 2
   * Fit Patients : CIRS (Cumulative Illness Rating Scale) less or equal 6
   * Life expectancy of more than 3 months

Note : Patients fulfilling the above inclusion criteria and presenting with the following features can also be included:

* patients with any rate of 17p deletion by FISH
* patients candidate for an allogeneic transplantation, provided these patients will be planned to receive the full BOMP treatment program and will have the final restaging assessment
* patients with fludarabine refractory disease
* patients with a prior diagnostic of CLL, at time of previous line(s) of treatment but who relapse without hyperlymphocytosis (lymphocytes < 5000/mm3) (lymphocytic lymphoma)
* prior monoclonal antibody (alemtuzumab or rituximab) exposure provided a washout period of 3 months before the start of the BOMP treatment.

Exclusion Criteria:

1. Untreated CLL
2. ECOG Performance Status > 2
3. Serious accompanying disorder or impaired organ function as indicated by:

   * Abnormal renal function with creatinine clearance < 40 ml/min calculated according to the formula of Cockcroft and Gault
   * Absolute neutrophils <1,000/mm3, platelets < 75000/mm3 (unless due to malignant B Cell involvement of the bone marrow and/or spleen enlargement)
   * Liver tests : total bilirubin >1.5 times UNL (unless due to CLL involvement of liver or a known history of Gilbert's disease), transaminases (ALAT, ASAT) and/or alkaline phosphatases >2.5 times UNL (unless due to CLL involvement of liver)
   * Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to study enrollment, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
   * Severe chronic obstructive pulmonary disease with hypoxemia or pulmonary diffusion capacity < 40 %
   * Uncontrolled diabetes mellitus,
   * Uncontrolled hypertension
   * History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
   * Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
4. CIRS (Cumulative Illness Rating Scale) > 6
5. Clinically significant auto-immune anemia [i.e. any drop in hemogolobin level related to an hemolytic autoimmune process attested by the following markers : elevated indirect bilirubin, elevated LDH, low haptoglobin levels, high reticulocytes count along with a positive direct anti-erythrocyte test (Coombs direct test)]
6. Transformation to an aggressive B-cell malignancy (e.g. diffuse large cell lymphoma, Hodgkin's lymphoma, or prolymphocytic leukaemia)
7. Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to start of therapy.
8. Prior autologous transplantation or allogeneic transplantation
9. Prior treatment with bendamustine and/or ofatumumab
10. Active second malignancy currently requiring treatment (except basal cell carcinoma, in situ cervix carcinoma and incidental prostate carcinoma). Subjects who have been free of malignancy for at least 5 years are eligible.
11. Known HIV-positivity
12. Positive serology for hepatitis B (HB) (except post vaccinale pattern) and/or for hepatitis C. Positive serology for HB is defined as a positive test for HBs antigen or for anti-HBc antibodies (regardless of HBsAb status).
13. Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment)
14. Simultaneous participation in another study protocol
15. Known hypersensitivity to the medications to be used specially to humanized monoclonal antibodies or any of the study drugs
16. Chronic or current bacterial, viral or fungal infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis
17. Any coexisting medical or psychological condition that would preclude participation in the required study procedures
18. Patient with mental deficiency preventing proper understanding of the requirements of treatment.
19. Pregnant or breastfeeding women.
20. Person major under law-control
21. Lactating women
22. Fertile male and female patients who cannot or do not wish to use an effective method of contraception, during and for 12 months after the final treatment used for the purposes of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Efficacy: Response rate according to IWCLL 2008 guidelines | 9 months
  Complete response rate (CR) at 6 cycles of BOMP according to IWCLL 2008 criteria Hallek 2008

SECONDARY OUTCOMES:
Tolerance and safety | 57 months
  Tolerance and safety of the BOMP regimen according to the CTC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Olivier TOURNILHAC, MD PD, Principal Investigator — French Innovative Leukemia Organisation; Sophie DE GUIBERT, MD PD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Tournilhac, Clermont-Ferrand, France

REFERENCES:
- See also: FILO Internet site — http://www.filo-leucemie.org